CLINICAL TRIAL: NCT03983096
Title: Pegylated Liposomal Doxorubicin or Epirubicin in Neoadjuvant or Adjuvant Chemotherapy for Breast Cancer: an Real-world, Multicenter, Case Control Study.
Brief Title: Pegylated Liposomal Doxorubicin or Epirubicin in Neoadjuvant or Adjuvant Chemotherapy for Breast Cancer.
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSPC-DMS-BC-13
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
Keywords: invasive breast cancer; neoadjuvant; adjuvant; Anthracycline
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- test group: Patients with invasive breast cancer diagnosed by menstrual histology in 2014-2018 and receiving neoadjuvant chemotherapy, or patients with invasive breast cancer diagnosed by menstrual histology in 2014-2016 and receiving adjuvant chemotherapy. That used Pegylated liposomal doxorubicin for treat.
- control group: Patients with invasive breast cancer diagnosed by menstrual histology in 2014-2018 and receiving neoadjuvant chemotherapy, or patients with invasive breast cancer diagnosed by menstrual histology in 2014-2016 and receiving adjuvant chemotherapy. That used epirubicin for treat.

SUMMARY:
Pegylated liposomal doxorubicin or epirubicin in neoadjuvant or adjuvant chemotherapy for breast cancer.

DETAILED DESCRIPTION:
This study is an real-world, multicenter, case control study about comparing pegylated liposomal doxorubicin Efficacy and safety of epirubicin in neoadjuvant and adjuvant chemotherapy for breast cancer. As this trial is a retrospective real-world study, investigator have given patients the dose of trial drugs based on real-world principles of diagnosis and treatment and their clinical experience. This trial only collects and analyzes patients' clinical medications, and does not interfere with patients' real-world diagnosis and treatment. A total of 1050 breast cancer patients are collecting from seven centers. 200 cases in neoadjuvant and 850 cases in adjuvant group. The follow-up examinations and assessment of the subjects were followed by real-world medical treatment routines and the visits were completed according to the routine of treatment. Related check and assessments and collect the following data: follow-up 3years or until the disease recurs (whichever occurs first). Adverse events: remission or stability of adverse events caused by follow-up to treatment in the adjuvant treatment group, follow-up for 3 years or until recurrence of the disease in the neoadjuvant treatment group (whichever first occurred).

ELIGIBILITY:
Inclusion Criteria:

1. Female;
2. Patients with invasive breast cancer diagnosed by menstrual histology in 2014-2018 and receiving neoadjuvant chemotherapy, or patients with invasive breast cancer diagnosed by menstrual histology in 2014-2016 and receiving adjuvant chemotherapy;
3. Chemotherapy regimen recommended by the guidelines for drugs containing anthracycline;
4. Patients whose chemotherapy regimen contains pegylated liposomal doxorubicin or epuroxorubicin;
5. Age :18 -70;
6. Patients with LVEF ≥ 50%.

Exclusion Criteria:

1. Patients with occult breast cancer.
2. Patients receiving two or more anthracyclines during neoadjuvant or adjuvant chemotherapy;
3. Patients who have previously received other chemotherapy regimens;
4. Patients with other malignant tumors in the past 5 years (except for cured cervical carcinoma in situ and basal cell carcinoma of the skin);
5. Patients complicated with severe infection and in need of treatment;
6. Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 1050 breast cancer patients were collected from seven centers. 200 cases in neoadjuvant and 850 cases in adjuvant group.
Sampling Method: Non-Probability Sample
Enrollment: 1213 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Pathological complete remission (pCR) | one year
  pCR was defned as no invasive cancer cells in any slices of the resected breast specimen.
Disease-free survival （DFS） | three years.
  The length of time after treatment during which no disease in found.

SECONDARY OUTCOMES:
Adverse event | three years
  Safety was assessed according to Common Terminology Criteria for Adverse Events version 4.0.
Breast conserving rate | one year
  Breast conserving operation rate.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Zhang, Pro., Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Jin Zhang, Tianjin, China